CLINICAL TRIAL: NCT01452776
Title: A Phase 3, Randomized, Single-Blind, Multicenter Study to Evaluate the Safety of TAK-438 (10 and 20 mg Once-daily) in a 52-week Maintenance Treatment in Patients With Healed Erosive Esophagitis (EE)
Brief Title: Long-Term Safety Study of TAK-438 in the Maintenance Treatment of Healed Erosive Esophagitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TAK-438/OCT-001; U1111-1123-9677 (Registry Identifier: WHO); JapicCTI-111615 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2011-09-16; First posted 2011-10-17 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Erosive Esophagitis
Keywords: Drug Therapy
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAK-438 10 mg QD (Experimental)
  Interventions: Drug: TAK-438
- TAK-438 20 mg QD (Experimental)
  Interventions: Drug: TAK-438

INTERVENTIONS:
Drug: TAK-438 — TAK-438 10 mg, tablets, orally, once daily for up to 52 weeks.
  Arms: TAK-438 10 mg QD
Drug: TAK-438 — TAK-438 20 mg, tablets, orally, once daily for up to 52 weeks.
  Arms: TAK-438 20 mg QD

SUMMARY:
The purpose of this study is to determine the safety of long term use of TAK-438, once daily (QD), for the maintenance treatment of healed erosive esophagitis.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have successfully completed the preceding phase 3 double-blind study (TAK-438/CCT-002: preceding study) and have endoscopically healed EE at Week 2, 4, or 8 in the preceding study.*

   * "Endoscopically healed EE" is defined as those participants who have endoscopically confirmed EE of Grade O as defined by the Los Angeles (LA) Classification Grading System.
2. Outpatient (including inpatient for examination)

Exclusion Criteria:

1. Participants with an esophagus-related complication (eosinophilic esophagitis, esophageal varices, scleroderma, viral or fungal infection, esophageal stenosis, etc.), a history of radiotherapy or cryotherapy of the esophagus, a caustic or physiochemical trauma (esophageal sclerotherapy, etc.). However, participants with Schatzki's ring (mucosal tissue ring around inferior esophageal sphincter) or Barrett's esophagus are allowed to be included.
2. Participants who have received surgery or treatment affecting gastroesophageal reflux (cardioplasty, dilation of esophageal stenosis [excluding Schatzki's ring], etc.), or who have a history of surgery of stomach or duodenum (excluding removal of benign polyp under endoscopy)
3. Participants who have acute upper gastrointestinal bleeding, gastric or duodenal ulcer (mucosal defect with white coating) within 30 days prior to Visit M-1 (initiation of study drug administration). However, participants with gastric or duodenal erosions are allowed to be included.
4. Participants with a previous or current history of Zollinger-Ellison syndrome, or other gastric acid hypersecretion disorder

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2011-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-emergent Adverse Events | 52 Weeks
  Treatment-emergent adverse events are defined as any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medicinal product reported from first dose of study drug through the last visit.

SECONDARY OUTCOMES:
Change from Baseline in Laboratory Values | Baseline and Week 52
Change from Baseline in Electrocardiograms | Baseline and Week 52
Change from Baseline in Vital Signs | Baseline and Week 52
Change from Baseline in Serum Gastrin | Baseline and Week 52
Change from Baseline in Pepsinogen I and II | Baseline and Week 52
Endoscopically confirmed recurrence rate of Erosive Esophagitis | 52 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Senior Manager, Study Director — Takeda
Locations (32):
- Japan (32):
  - Nagoya, Aichi-ken
  - Abiko-shi, Chiba
  - Fukuoka, Fukuoka
  - Itoshima-shi, Fukuoka
  - Kurume-shi, Fukuoka
  - Onga-gun, Fukuoka
  - Gifu, Gifu
  - Annaka-shi, Gunma
  - Aki-gun, Hiroshima
  - Hiroshima, Hiroshima
  - Sapporo, Hokkaido
  - Amagasaki-shi, Hyōgo
  - Kobe, Hyōgo
  - Takarazuka-shi, Hyōgo
  - Sakaide-shi, Kagawa-ken
  - Yokohama, Kanagawa
  - Kochi, Kochi
  - Susaki-shi, Kochi
  - Kumamoto, Kumamoto
  - Kyoto, Kyoto
  - Nagasaki, Nagasaki
  - Ōita, Oita Prefecture
  - Okayama, Okayama-ken
  - Fuziidera-shi, Osaka
  - Shizuoka, Shizuoka
  - Otawara-shi, Tochigi
  - Chiyoda-ku, Tokyo
  - Chuo-ku, Tokyo
  - Nakano-ku, Tokyo
  - Ōta-ku, Tokyo
  - Setagaya-ku, Tokyo
  - Yamagata, Yamagata